CLINICAL TRIAL: NCT03689023
Title: Health Promotion and Cardiovascular Risk Reduction Among People With Spinal Cord Injury: Physical Activity, Healthy Diet and Maintenance After Discharge.
Brief Title: Health Promotion and Cardiovascular Risk Reduction Among People With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Metropolitan University College (Other)
Responsible Party: Principal Investigator, Nicolaj Jersild Holm, Principal investigator, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Primary study
Record Dates: First submitted 2018-08-01; First posted 2018-09-28 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Spinal Cord Injuries
Keywords: Cardiovascular Diseases; Health Promotion
MeSH Terms: conditions — Spinal Cord Injuries; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A controlled multimodal intervention (Experimental): A uniform and systematic patient education about cardiovascular risk factors, physical activity and a healthy diet lifestyle starting early in the primary rehabilitation process with 6 months of follow up.
  Interventions: Other: A controlled multimodal intervention

INTERVENTIONS:
Other: A controlled multimodal intervention — The intervention is interdisciplinary, multimodal and patient activating and uses the existing setting and work flows at the Clinic as well as new interventions, ensuring that the patients receive education about cardiovascular risk factors, physical activity and healthy diet through a systematic approach including targeted patient education

SUMMARY:
This study is a controlled pragmatic implementation study in clinical practice, with a primary focus on cardiovascular risk reduction through adherence to behavioral interventions related to physical activity and healthy diet.The intervention is interdisciplinary, multimodal and patient activating and uses the existing setting and work flows at the clinic, ensuring that the patients receive education about cardiovascular risk factors, physical activity and healthy diet through a systematic approach including targeted patient education.

DETAILED DESCRIPTION:
This clinical intervention study will investigate the effectiveness of a uniform and systematic institutional strategy incorporating targeted strategic patient education about cardiovascular risk factors, physical activity and a healthy diet lifestyle starting early in the primary rehabilitation process with 6 months of follow up compared to a historic control group. Test - retest reliability of four different VO2 peak tests and a multi sensor accelerometer respectively will be assessed as well.

ELIGIBILITY:
Inclusion Criteria:

* All newly injured patients (within the last 12 months) with Spinal Cord Injury admitted at Clinic for Spinal Cord Injuries, Rigshospitalet.

Exclusion Criteria:

* Insufficient skills in Danish language
* Reduced mental function that prevents reading and answering the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
VO2peak | Assessing change from admission to discharge in average 4-6 months after admission and follow up 6 months after discharge
  Measures peak oxygen consumption in ml/kg/min

SECONDARY OUTCOMES:
Body Mass Index | At admission
  Defined as a person's weight in kilograms divided by the square of the person's height in metres (kg/m2
Body Mass Index | At discharge in average 4-6 months after admission
  Defined as a person's weight in kilograms divided by the square of the person's height in metres (kg/m2
Body Mass Index | At follow up 6 months after discharge
  Defined as a person's weight in kilograms divided by the square of the person's height in metres (kg/m2
International Standards for Neurological Classification of Spinal Cord Injury | At admission
  The classification tool involves a sensory and motor examination to determine the neurological level of the injury and whether the injury is complete or incomplete. It defines neurological level as the most caudal level at which sensory and motor function are intact. The completeness of the injury is graded from A to E according to the American Spinal Injury Assosciation Impairment Scale (AIS). Grade A indicates a worse score and E indicates a better score
International Standards for Neurological Classification of Spinal Cord Injury | At discharge in average 4-6 months after admission
  The classification tool involves a sensory and motor examination to determine the neurological level of the injury and whether the injury is complete or incomplete. It defines neurological level as the most caudal level at which sensory and motor function are intact. The completeness of the injury is graded from A to E according to the American Spinal Injury Assosciation Impairment Scale (AIS). Grade A indicates a worse score and E indicates a better score
International Standards for Neurological Classification of Spinal Cord Injury | At follow up 6 months after discharge
  The classification tool involves a sensory and motor examination to determine the neurological level of the injury and whether the injury is complete or incomplete. It defines neurological level as the most caudal level at which sensory and motor function are intact. The completeness of the injury is graded from A to E according to the American Spinal Injury Assosciation Impairment Scale (AIS). Grade A indicates a worse score and E indicates a better score
Leisure Time Physical Activity Questionnaire for people with Spinal Cord Injury | At admission
  Questionnaire concerning the amount of leisure time physical activity the past 7 days. The patient describes how many of the last 7 days and for how many minutes he/she has been physical active and also the intensity of the activity described as mild, moderate or vigorous. Higher values related to days, minutes and intensity represent a better outcome and lower values represent a worse outcome.On the scale related to days, 0 is a minimum score and 7 is a maximum score.
Leisure Time Physical Activity Questionnaire for people with Spinal Cord Injury | At discharge in average 4-6 months after admission
  Questionnaire concerning the amount of leisure time physical activity the past 7 days. The patient describes how many of the last 7 days and for how many minutes he/she has been physical active and also the intensity of the activity described as mild, moderate or vigorous. Higher values related to days, minutes and intensity represent a better outcome and lower values represent a worse outcome.On the scale related to days, 0 is a minimum score and 7 is a maximum score.
Leisure Time Physical Activity Questionnaire for people with Spinal Cord Injury | At follow up 6 months after discharge
  Questionnaire concerning the amount of leisure time physical activity the past 7 days. The patient describes how many of the last 7 days and for how many minutes he/she has been physical active and also the intensity of the activity described as mild, moderate or vigorous. Higher values related to days, minutes and intensity represent a better outcome and lower values represent a worse outcome.On the scale related to days, 0 is a minimum score and 7 is a maximum score.
The Exercise Self Efficacy Scale for people with Spinal Cord Injury | At admission
  A questionnaire with a 4-point rating scale describing how confident persons with spinal cord injury are with regard to carrying out regular physical activities and exercise. The questionnaire consists of 10 items with corresponding response options on a 4-point Likert scale (1-not at all true, 4-always true) with 1 indicating a worse score and 4 indicating a better score. The total score is derived by summing the scores for the individual items with a possible score range from 10 to 40.
The Exercise Self Efficacy Scale for people with Spinal Cord Injury | At discharge in average 4-6 months after admission
  A questionnaire with a 4-point rating scale describing how confident persons with spinal cord injury are with regard to carrying out regular physical activities and exercise. The questionnaire consists of 10 items with corresponding response options on a 4-point Likert scale (1-not at all true, 4-always true) with 1 indicating a worse score and 4 indicating a better score. The total score is derived by summing the scores for the individual items with a possible score range from 10 to 40.
The Exercise Self Efficacy Scale for people with Spinal Cord Injury | At follow up 6 months after discharge
  A questionnaire with a 4-point rating scale describing how confident persons with spinal cord injury are with regard to carrying out regular physical activities and exercise. The questionnaire consists of 10 items with corresponding response options on a 4-point Likert scale (1-not at all true, 4-always true) with 1 indicating a worse score and 4 indicating a better score. The total score is derived by summing the scores for the individual items with a possible score range from 10 to 40.
Dual energy x-ray absorbtiometry (Dexa) | At admission
  Assessment of lean body mass percentage
Dual energy x-ray absorbtiometry (Dexa) | At follow up 6 months after discharge
  Assessment of lean body mass percentage
Blood pressure | At admission
  Assessment of both systolic and diastolic blood pressure in mm/ Hg
Blood pressure | At discharge in average 4-6 months after admission
  Assessment of both systolic and diastolic blood pressure in mm/ Hg
Blood pressure | At follow up 6 months after discharge
  Assessment of both systolic and diastolic blood pressure in mm/ Hg
The 9-item Shared Decision Making Questionnaire (SDM-Q-9) | At discharge in average 4-6 months after admission
  The SDM-Q-9 is a questionnaire describing the process of Shared Decision Making between health care professionals and the patient from the patient's perspective and consists of nine statements, which can be rated on a six-point scale from ''completely disagree'' (0) being the worse score to ''completely agree'' (5) being the better score. Summing up all items leads to a raw total score between 0 and 45.
Triglycerides | At admission
  Assessment of plasma triglycerides in mmol/l
Triglycerides | At discharge in average 4-6 months after admission
  Assessment of plasma triglycerides in mmol/l
Triglycerides | At follow up 6 months after discharge
  Assessment of plasma triglycerides in mmol/l
Cholesterol | At admission
  Assessment of cholesterol in mmol/l
Cholesterol | At discharge in average 4-6 months after admission
  Assessment of cholesterol in mmol/l
Cholesterol | At follow up 6 months after discharge
  Assessment of cholesterol in mmol/l
HemoglobinA1c | At admission
  A marker for carbohydrate metabolism measured in mmol/mol
HemoglobinA1c | At discharge in average 4-6 months after admission
  A marker for carbohydrate metabolism measured in mmol/mol
HemoglobinA1c | At follow up 6 months after discharge
  A marker for carbohydrate metabolism measured in mmol/mol
C - reactive protein (CRP) | At admission
  A clinical biomarker that signposts non-specific inflammation measured in Mg/L
C - reactive protein (CRP) | At discharge in average 4-6 months after admission
  A clinical biomarker that signposts non-specific inflammation measured in Mg/L
C - reactive protein (CRP) | At follow up 6 months after discharge
  A clinical biomarker that signposts non-specific inflammation measured in Mg/L

OTHER OUTCOMES:
Spinal Cord Injury Independence Measure III | At admission
  The SCIM is composed of 19 items that assess 3 domains.1 Self-care (6 items, scores range from 0-20). 2 Respiration and sphincter management (4 items, scores range from 0-40). 3 Mobility (9 items, scores range from 0-40). The total SCIM scores range from 0 to 100.
Spinal Cord Injury Independence Measure III | At discharge in average 4-6 months after admission
  The SCIM is composed of 19 items that assess 3 domains.1 Self-care (6 items, scores range from 0-20). 2 Respiration and sphincter management (4 items, scores range from 0-40). 3 Mobility (9 items, scores range from 0-40). The total SCIM scores range from 0 to 100.
Spinal Cord Injury Independence Measure III | At follow up 6 months after discharge
  The SCIM is composed of 19 items that assess 3 domains.1 Self-care (6 items, scores range from 0-20). 2 Respiration and sphincter management (4 items, scores range from 0-40). 3 Mobility (9 items, scores range from 0-40). The total SCIM scores range from 0 to 100.
Patient Health Questionnaire- 2 | At admission
  The PHQ-2, comprising the first 2 items of the PHQ-9, inquires about the degree to which an individual has experienced depressed mood and anhedonia over the past two weeks Score range is from from 0- 3, with 0 indicating a better score. Total score ranges from 0 (minimum score to 6 (maximum score), with 0 indicating a better score and with a cut-off score of 3 as the cut point for screening purposes.
Patient Health Questionnaire- 2 | At discharge in average 4-6 months after admission
  The PHQ-2, comprising the first 2 items of the PHQ-9, inquires about the degree to which an individual has experienced depressed mood and anhedonia over the past two weeks Score range is from from 0- 3, with 0 indicating a better score. Total score ranges from 0 (minimum score to 6 (maximum score), with 0 indicating a better score and with a cut-off score of 3 as the cut point for screening purposes.
Patient Health Questionnaire- 2 | At follow up 6 months after discharge
  The PHQ-2, comprising the first 2 items of the PHQ-9, inquires about the degree to which an individual has experienced depressed mood and anhedonia over the past two weeks Score range is from from 0- 3, with 0 indicating a better score. Total score ranges from 0 (minimum score to 6 (maximum score), with 0 indicating a better score and with a cut-off score of 3 as the cut point for screening purposes.
The International SCI Quality of Life Basic Data Set | At admission
  Consists of three questions scored on a scale of 0-10 regarding general quality of life, physical health and satisfaction with psychological Health. 0 indicates a worse score and 10 indicates a better score.
The International SCI Quality of Life Basic Data Set | At discharge in average 4-6 months after admission
  Consists of three questions scored on a scale of 0-10 regarding general quality of life, physical health and satisfaction with psychological Health. 0 indicates a worse score and 10 indicates a better score.
The International SCI Quality of Life Basic Data Set | At follow up 6 months after discharge
  Consists of three questions scored on a scale of 0-10 regarding general quality of life, physical health and satisfaction with psychological Health. 0 indicates a worse score and 10 indicates a better score.
Objective physical activity (accelerometry) | At admission
  Is measured with a multisensor device (Actiheart®) measuring physical activity energy expenditure in kcal/min.
Objective physical activity (accelerometry) | At follow up 6 months after discharge
  Is measured with a multisensor device (Actiheart®) measuring physical activity energy expenditure in kcal/min..
Objective physical activity (accelerometry) | At discharge in average 4-6 months after admission
  Is measured with a multisensor device (Actiheart®) measuring physical activity energy expenditure in kcal/min..
The Nordic monitoring of diet, physical activity and overweight (NORMON) | At admission
  The questionnaire Is used to measure the course in dietary habits and explores how often 16 food indicators are consumed. The food indicators are chosen in a way that reflects the diets nutritional quality. An association between the frequency of food indicator intake and the overall nutritional value of the diet is present. Several of the chosen food indicators are recommended in the national nutritional recommendations.
The Nordic monitoring of diet, physical activity and overweight (NORMON) | At discharge in average 4-6 months after admission
  The questionnaire Is used to measure the course in dietary habits and explores how often 16 food indicators are consumed. The food indicators are chosen in a way that reflects the diets nutritional quality. An association between the frequency of food indicator intake and the overall nutritional value of the diet is present. Several of the chosen food indicators are recommended in the national nutritional recommendations.
The Nordic monitoring of diet, physical activity and overweight (NORMON) | At follow up 6 months after discharge
  The questionnaire Is used to measure the course in dietary habits and explores how often 16 food indicators are consumed. The food indicators are chosen in a way that reflects the diets nutritional quality. An association between the frequency of food indicator intake and the overall nutritional value of the diet is present. Several of the chosen food indicators are recommended in the national nutritional recommendations.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for Spinal Cord Injuries, Rigshopitalet, Hornbæk, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holm NJ, Moller T, Adamsen L, Dalsgaard LT, Biering-Sorensen F, Schou LH. Health promotion and cardiovascular risk reduction in people with spinal cord injury: physical activity, healthy diet and maintenance after discharge- protocol for a prospective national cohort study and a preintervention- postintervention study. BMJ Open. 2019 Dec 31;9(12):e030310. doi: 10.1136/bmjopen-2019-030310. PMID 31892644

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/23/NCT03689023/Prot_SAP_001.pdf